CLINICAL TRIAL: NCT02007954
Title: Doxorubicin-eluting LC Bead M1 for Patients With Hepatocellular Carcinoma (DEBDOX)
Brief Title: Doxorubicin-eluting LC Bead M1 for Patients With Hepatocellular Carcinoma
Acronym: DEBDOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1306; NA_00077927 (Other: JHMIRB)
Record Dates: First submitted 2013-11-21; First posted 2013-12-11 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2014-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DEBDOX (Experimental)
  Interventions: Device: DEBDOX

INTERVENTIONS:
Device: DEBDOX — DEBDOX, loaded with doxorubicin, is a device that utilizes beads in place of lipiodol to deliver the chemotherapy into the liver tumor. The device allows for continuous elution of doxorubicin into the liver tumor tissue. The advantages of this method of delivery in comparison to conventional TACE are that the beads are able to deliver a greater volume and concentration of the drugs to the tumor because of their unique ability to elute the drug over a period of several days. As a result of this unique delivery, systemic toxicity is significantly reduced. The potential advantages of the smaller beads are deeper penetration into the tumor bed, while avoiding premature proximal occlusion of vessels feeding the tumor, and more consistent dosing. These properties translate into greater potency of therapy and potentially improved patient survival.

SUMMARY:
The purpose of this study is to determine the feasibility and safety of using small beads (70-150 micron in place of 100-300 micron) to deliver chemotherapy into the liver to treat patients with hepatocellular carcinoma (HCC). The beads (LC-Bead M1) will be loaded with doxorubicin (DEBDOX-M1), and used to administer transarterial chemoembolization (TACE) DEBDOX, loaded with doxorubicin, is a device that utilizes tiny beads (70-150 microns) to deliver chemotherapy agents into liver tumor(s) via the hepatic artery. This device allows for continuous release of doxorubicin into the liver tumor tissue(s) causing necrosis of the targeted tumor(s). The potential advantages of the smaller beads are deeper penetration into the tumor bed, while avoiding premature proximal occlusion of vessels feeding the tumor, and more consistent dosing. Response to therapy will be evaluated monthly by clinic visits and blood tests (to include assessment of liver function and tumor markers) and by imaging (usually MRIs) every 1-2 months. Patients will be on study for 6 months after which they will be exited from the study and followed for survival. Once exited from the study they will continue to be eligible to receive the smaller beads (DEBDOX), should it be recommended.

ELIGIBILITY:
INCLUSION CRITERIA:

1. The patient has preserved liver function (Child-Pugh A-B class) without significant liver decompensation.
2. The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at study entry.
3. The patient is age 18 years or older.
4. The patient has a life expectancy of > 12 weeks.
5. The patient has measurable or evaluable disease that will be directly treated with intrahepatic therapy (as defined by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).
6. The patient has adequate hematologic function as defined by the following criteria:

   * An absolute neutrophil count (ANC) ≥ 1500/micro L,
   * Hemoglobin ≥ 9.5 g/dL, and a
   * Platelet count ≥ 50,000/micro L.
7. The patient has adequate hepatic function, as defined by the following criteria:

   * Total bilirubin </= 3.0 mg/dL
   * Aspartate transaminase (AST) and alanine transaminase (ALT) </= 8 x the upper limit of normal (ULN).
8. The patient has adequate renal function, as defined by the following criteria:

   * Serum creatinine </= 2.0 x the institutional ULN
9. The patient has a baseline international normalized ratio (INR) < 1.5.
10. The patient, if a woman of childbearing potential, has a negative pregnancy test.
11. The patient is able to give written informed consent.
12. The patient is willing and able to comply with study procedures, scheduled visits, and treatment plans.
13. Patients with early stage HCC may be included in the protocol to receive DEBDOX-M1 prior to resection

EXCLUSION CRITERIA:

1. The patient has a history of another primary cancer (ie, a primary cancer not associated with the patient's current liver tumor), with the exception of (a) curatively resected nonmelanomatous skin cancer; (b) curatively treated cervical carcinoma in situ; or (c) other primary solid tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years prior to enrollment (date of informed consent).
2. The patient is receiving concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemoembolization, targeted therapy, or an investigational agent.
3. The patient has extrahepatic, metastatic, symptomatic HCC. Enlarged reactive lymph nodes, or indeterminate lesions, such as lung nodules are acceptable.
4. The patient's tumor has replaced >70% of the liver volume.
5. The patient has clinically significant ascites. Trace ascites on imaging is acceptable.
6. Marco-shunting noted on the hepatic angiogram.
7. The patient has untreatable bleeding diathesis.
8. The patient has complete main portal vein thrombosis with reversal of flow.
9. The patient has a left ventricle ejection fraction of less than 45%.
10. The patient has evidence of clinically significant peripheral vascular disease.
11. The patient has clinically significant or symptomatic extrahepatic disease, for example, an uncontrolled inter-current illness including, but not limited to:

    * Ongoing or active infection requiring parenteral antibiotics
    * Symptomatic congestive heart failure (class II to IV of the New York Heart Association classification for heart disease)
    * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
    * Uncontrolled hypertension (systolic blood pressure > 150 mmHg, diastolic blood pressure > 90 mmHg, found on 2 consecutive measurements separated by a 1-week period despite adequate medical support)
    * Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [NCI-CTCAE Grade 3] or asymptomatic sustained ventricular tachycardia)
    * Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements
12. There is evidence of substance abuse or medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results.
13. The patient is pregnant or breast-feeding.
14. The patient is allergic to contrast media that cannot be readily prevented with premedication or managed.
15. The patient has extra-hepatic, metastatic, and symptomatic HCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08-11 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Geschwind, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled patients diagnosed with unresectable hepatocellular carcinoma without prior locoregional therapy or concurrent anticancer therapy. Patients were enrolled from February 2014 to January 2015, with the last patient completing follow-up in August 2015.
Period: Overall Study
Arm/Group | DEBDOX
Started | 24 (A total of 32 participants were consented, with 8 patients screened out prior to treatment.)
Completed First TACE (Number of patients who completed the first treatment on protocol and included in analysis) | 24
Completed First Clinical and Imaging (Participants completing this milestone will be analyzed for image response outcomes) | 23 (1 patient exited prior to first imaging follow-up due to unrelated serious adverse event and death)
Completed (Participants who have completed all 6 months of treatment on trial) | 17
Not Completed | 7
Not completed — Received liver transplant | 3
Not completed — Switch in treatment modality | 2
Not completed — Disease progression and unrelated AE | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | DEBDOX
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 62.5 [35 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Out of 24 enrolled participants, 23 participants identified as non-Hispanic and 1 did not elect to reveal their ethnicity. From the 24 participants, 15 were white, 7 were black or African American, 1 was Asian, and 1 was unknown.
  Participants
    Non-Hispanic: number analyzed (Participants) | 23
    Non-Hispanic: White | 15
    Non-Hispanic: African American | 7
    Non-Hispanic: Asian | 1
    Non-Hispanic: Unknown | 0
    Unknown: number analyzed (Participants) | 1
    Unknown: White | 0
    Unknown: African American | 0
    Unknown: Asian | 0
    Unknown: Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Success of DEBDOX-M1 Procedure as a Measure of Feasibility
Description: Feasibility is defined as achieving an acceptable level of technical success in the use of DEBDOX-M1 beads treating hepatic lesions in patients with hepatocellular carcinoma.
Time Frame: 6 months
Population: The 24 patients received a total of 50 DEBDOX-M1 TACE procedures.
Measure: Number; unit: percentage of successful treatments
Units Other Than Participants: DEBDOX-M1 treatments
Arm/Group | DEBDOX
Number analyzed (Participants) | 24
Number analyzed (DEBDOX-M1 treatments) | 50
percentage of successful treatments | 100

2. Primary Outcome: Collection of Adverse Events Related to Study Device as a Measure of Safety
Description: For safety, all toxicities assessed as being at least possibly related will be analyzed by descriptive statistics to show type, grade (NCI Common Toxicity Criteria v.4 toxicity criteria), frequency and time from DEBDOX-M1TACE.
Time Frame: 1 month
Population: 30-day toxicity report of device-related adverse events for all 24 patients with classification and grading based on CTCAE v4.0.
Measure: Number; unit: Adverse Events
Arm/Group | DEBDOX
Number analyzed (Participants) | 24
Adverse Events
  Hypertension | 6
  Anorexia | 4
  Fatigue | 2
  Fever | 2
  Weight loss | 1
  Weight gain | 1
  Insomnia | 1
  Hyperglycemia | 5
  Hypoglycemia | 1
  Ascites | 1
  Diarrhea | 2
  Constipation | 1
  Gas | 1
  Nausea/Vomiting | 1
  Groin hematoma | 1
  Hyperbilirubinemia | 2
  Hypoalbuminemia | 1
  Cellulitis | 1
  Headache | 2
  Confusion | 1
  Abdominal non-specific pain | 2
  Pain - general | 1
  Pain - right shoulder | 1
  Hypercreatininemia | 1
  Hypokalemia | 1
  Hyponatremia | 3
  Grade 3 Elevated Transaminase | 1
  Hypoxia | 1
  Cardiac arrest | 1
  Total Grade 1-2 adverse events | 46
  Total Grade 3 or higher adverse events | 3

3. Secondary Outcome: Efficacy - Tumor Response by EASL
Description: Efficacy as assessed by radiographic tumor response using EASL amendment at baseline and at 1 month imaging following TACE treatments.
  Complete Response (CR): Achieving 100% tumor necrosis of lesions targeted by DEBDOX-M1. Baseline degree of tumor enhancement used as a reference.
  Partial Response (PR): Demonstrating greater than 50% tumor necrosis in lesions targeted by DEBDOX-M1.
  Stable Disease (SD): Not meeting requirements for CR or PR and not demonstrating evidence of progression of lesions targeted by DEBDOX-M1.
  Progressive Disease (PD): Reappearance of or increased tumor enhancement greater than 25% in lesions previously targeted by DEBDOX-M1.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | DEBDOX
Number analyzed (Participants) | 23
Participants
  Complete Response | 5
  Partial Response | 5
  Stable Disease | 10
  Progressive Disease | 3
  Objective response (CR + PR) | 10
  Disease control rate (CR + PR + SD) | 20

4. Secondary Outcome: Efficacy - Tumor Response by qEASL
Description: Efficacy as assessed by radiographic tumor response using qEASL at baseline and at 1-month imaging following TACE treatments.
  Complete Response (CR): Disappearance of any intratumoral arterial enhancement in all target lesions.
  Partial Response (PR): At least a 65% decrease in the sum of enhancing tissue volume of the lesions.
  Stable Disease (SD): Any cases that do not qualify for complete response, partial response, or progressive disease.
  Progressive Disease (PD): an increase of at least 73% in the sum of enhancing tissue volume of the lesions.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | DEBDOX
Number analyzed (Participants) | 23
Participants
  Complete Response | 5
  Partial Response | 4
  Stable Disease | 13
  Progressive Disease | 1
  Objective response (CR + PR) | 9
  Disease control rate (CR + PR + SD) | 22

5. Secondary Outcome: Efficacy - Tumor Response by mRECIST
Description: Efficacy as assessed by radiographic tumor response using modified RECIST (mRECIST) criteria at baseline and at 1-month imaging following TACE treatments.
  Complete Response (CR): Disappearance of any intratumoral arterial enhancement in all target lesions Partial Response (PR): At least 30% decrease in the sum of diameters of viable target lesions, taking as reference the baseline sum of the diameters of target lesions Progressive Disease (PD): At least 20% increase in the sum of diameters of viable target lesions, taking as reference the smallest sum of diameters of viable target lesions since treatment started Stable Disease (SD): Any cases that do not qualify for either PR or PD.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | DEBDOX
Number analyzed (Participants) | 23
Participants
  Complete Response | 5
  Partial Response | 5
  Stable Disease | 11
  Progressive Disease | 2
  Objective response (CR + PR) | 10
  Disease control rate (CR + PR + SD) | 21

6. Secondary Outcome: Efficacy - Number of Patients Downstaged or Bridged to Surgical Interventions
Description: The number of patients who underwent a liver transplantation following treatment on this protocol.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DEBDOX
Number analyzed (Participants) | 24
Participants | 6

7. Secondary Outcome: AFP Tumor Marker Pre- and Post-treatment
Description: The change in alpha-fetoprotein tumor marker levels pre- and post-treatment with one DEBDOX-M1 TACE procedure.
Time Frame: 1 month
Population: 23 out of 24 patients analyzed due to one patient not completing AFP post-TACE.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | DEBDOX
Number analyzed (Participants) | 23
ng/mL
  Pre-M1 TACE | 289.7 [1.8 to 4152]
  Post-M1 TACE | 145.4 [1.3 to 1706.5]
Statistical Analysis 1: Comparison: DEBDOX; Shapiro-Wilk test was run for normality. Baseline and follow-up AFP compared using two-tailed Student's t-test; Test type: Other; p = .01, t-test, 2 sided — P-values < 0.05 considered statistically significant

8. Other Pre Specified Outcome: Exploratory Endpoint - Pharmacokinetic (PK) Profile of Doxorubicin and Doxorubicinol Post DEBDOX-M1 TACE
Description: PK analysis of doxorubicin and its metabolite doxorubicinol post DEBDOX-M1 in the first 10 patients enrolled on protocol including peak plasma concentration (Cmax).
  Time points assessed in protocol were pre-dose, and then 5min, 20min, 40min, 1hr, 2hr, and 24hr post administration of 50-100mg doxorubicin.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DEBDOX
Number analyzed (Participants) | 10
ng/mL | 139.9 (98.2)

9. Other Pre Specified Outcome: Exploratory Endpoint - Total Drug Exposure Over Time (AUC) of Doxorubicin and Doxorubicinol Post TACE
Description: Total drug exposure over time (AUC) of doxorubicin and its metabolite doxorubicinol post DEBDOX in the first 10 patients enrolled on protocol. Time points assessed in protocol were pre-dose, and then 5min, 20min, 40min, 1hr, 2hr, and 24hr post administration of 50-100mg doxorubicin..
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DEBDOX
Number analyzed (Participants) | 10
ng*h/mL | 327 (366)

10. Other Pre Specified Outcome: Exploratory Endpoint - Tmax of Doxorubicin and Doxorubicinol Post DEBDOX-M1 TACE
Description: Time taken to reach maximum concentration (Tmax) of doxorubicin and its metabolite doxorubicinol post DEBDOX-M1 in the first 10 patients enrolled on protocol. Time points assessed in protocol were pre-dose, and then 5min, 20min, 40min, 1hr, 2hr, and 24hr post administration of 50-100mg doxorubicin..
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DEBDOX
Number analyzed (Participants) | 10
minutes | 6.6 (3.6)

ADVERSE EVENTS:
Time Frame: Adverse events collected over the participant's duration on study (6 months)
Arm/Group | DEBDOX
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEBDOX (N=24)
Cardiac arrest (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEBDOX (N=24)
Abdominal pain (Gastrointestinal disorders) | 10 (12)
Anemia (Blood and lymphatic system disorders) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Ascites (Gastrointestinal disorders) | 3 (4)
Intrahepatic biloma (Hepatobiliary disorders) | 1 (1)
Pain (General disorders) | 7 (9)
Skin abscess (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 10 (12)
Aspartate aminotransferase (Investigations) | 9 (10)
INR increased (Investigations) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 13 (19)
Fever (General disorders) | 4 (4)
Flu like symptoms (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Hematoma (Vascular disorders) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 11 (14)
Creatinine increased (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (22)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 14 (16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (18)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (8)
Hemoglobin increased (Investigations) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
White blood cell decreased (Investigations) | 7 (12)
Lymphocyte count decreased (Investigations) | 11 (14)
Malaise (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6)
Neutrophil count decreased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 5 (5)
Upper respiratory infection (Infections and infestations) | 1 (1)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes